CLINICAL TRIAL: NCT03057587
Title: The Newborn Project: A Prospective Observational Study Examining the Oxygenation of Brain Tissue During General Anesthesia Using Near Infrared Spectroscopy Technology
Brief Title: The Newborn Project: Examining the Oxygenation of Brain Tissue During General Anesthesia
Status: Withdrawn | Type: Observational
Why Stopped: The research never began.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Mary Ellen McCann, MD, MPH, Boston Children's Hospital
Other Study IDs: IRB-P00021194
Record Dates: First submitted 2017-02-15; First posted 2017-02-20 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NIRS Monitoring: A NIRS sensor will be placed on the forehead of the patient upon entry to the operating room and will remain on, as tolerated, for the duration of surgery
  Interventions: Device: NIRS Monitoring

INTERVENTIONS:
Device: NIRS Monitoring — NIRS data will be collected throughout the surgery

SUMMARY:
This study will be an observational, prospective trial that will measure the cerebral oxygenation of infants scheduled to undergo general anesthesia at Boston Children's Hospital.

DETAILED DESCRIPTION:
Data will be collected from the Near Infrared Spectroscopy (NIRS) monitor and the patient's medical record. When the NIRS sensor is attached to the patient's forehead the oxygenation of brain tissue will be continuously monitored. All other information will be routinely recorded as standard clinical care and this information will be obtained from the patient's medical record. The NIRS monitor data will by time synched to the anesthesia record and downloaded to a secured password protected file.

In the post-operative period, patient data will be collected including: 1) any skin findings related to the placement of the NIRS or pulse oximetry probes 2) any unanticipated need for hemodynamic support, 3) laboratory values including hemoglobin levels, electrolytes, and blood gases, 4) new neurological findings (seizures etc.)

ELIGIBILITY:
Inclusion Criteria:

* Children less than 6 months of age
* Undergoing a scheduled or emergent procedure with anesthesia at Boston Children's Hospital

Exclusion Criteria:

* Placement of NIRS sensor that will interfere with surgery
* Child has an allergy to medical grade adhesives or pre-existing skin irritation at the sensor site
* Scheduled for a cardiac procedure
* Patient's care team or patient's family declines participation
* American Society of Anesthesiologists (ASA) criteria of IV or greater
* Infants who are being treated with sympathomimetic medications intraoperatively

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants scheduled to undergo general anesthesia at Boston Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-04-27 (Actual)

PRIMARY OUTCOMES:
Cerebral Oxygenation | Intraoperative period
  Determine what factors are correlated with changes in the cerebral oxygenation

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ellen McCann, MD, MPH, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Graaff JC, Pasma W, van Buuren S, Duijghuisen JJ, Nafiu OO, Kheterpal S, van Klei WA. Reference Values for Noninvasive Blood Pressure in Children during Anesthesia: A Multicentered Retrospective Observational Cohort Study. Anesthesiology. 2016 Nov;125(5):904-913. doi: 10.1097/ALN.0000000000001310. PMID 27606930
- [Background] Aly SA, Zurakowski D, Glass P, Skurow-Todd K, Jonas RA, Donofrio MT. Cerebral tissue oxygenation index and lactate at 24 hours postoperative predict survival and neurodevelopmental outcome after neonatal cardiac surgery. Congenit Heart Dis. 2017 Mar;12(2):188-195. doi: 10.1111/chd.12426. Epub 2016 Nov 10. PMID 27862979
- [Background] Razlevice I, Rugyte DC, Strumylaite L, Macas A. Assessment of risk factors for cerebral oxygen desaturation during neonatal and infant general anesthesia: an observational, prospective study. BMC Anesthesiol. 2016 Oct 28;16(1):107. doi: 10.1186/s12871-016-0274-2. PMID 27793105
- [Background] Michelet D, Arslan O, Hilly J, Mangalsuren N, Brasher C, Grace R, Bonnard A, Malbezin S, Nivoche Y, Dahmani S. Intraoperative changes in blood pressure associated with cerebral desaturation in infants. Paediatr Anaesth. 2015 Jul;25(7):681-8. doi: 10.1111/pan.12671. Epub 2015 Apr 30. PMID 25929346